CLINICAL TRIAL: NCT01762592
Title: A Study of Iodine (124I) Girentuximab PET/CT Scan for the Detection of Clear Cell Renal Cell Carcinoma in Patients With Indeterminate cT1 Renal Masses
Brief Title: REDECT 2: REnal Masses: Pivotal Trial to DEteCT Clear Cell Renal Cell Carcinoma With PET/CT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: new sponsor
Sponsor: Heidelberg Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WX/20-002
Record Dates: First submitted 2012-12-19; First posted 2013-01-07 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Renal Cell Carcinoma; Kidney Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Iodine; G250 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Iodine (124I) Girentuximab (Experimental): Single infusion of radio labeled antibody: 30 mL will be infused using an infusion pump at a rate of 2mL/min over 15 minutes on study day 0.
  Interventions: Drug: Iodine (124I) Girentuximab

INTERVENTIONS:
Drug: Iodine (124I) Girentuximab — i.v.
  Other Names: 124I-cG250

SUMMARY:
Study WX-20-002 will confirm diagnostic efficacy and safety of a PET/CT scan using Iodine (124I) Girentuximab performed during the diagnostic work-up in patients with indeterminate cT1-renal masses.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age.
2. Presence of indeterminate cT1 renal mass by screening CT with and without contrast or MRI with and without contrast (MRI only if CT is contra-indicated).
3. Negative serum pregnancy test; to be performed on female patients of childbearing potential within 24 hours prior to receiving investigational product.
4. Recovered from toxicity of any prior therapy to grade 1 or better.
5. Able to take oral medication (KI).
6. Written informed consent available.

Exclusion Criteria:

1. Renal mass known to be a metastasis of another primary tumor.
2. Known histology of renal mass (e.g. by biopsy).
3. Active non-renal malignancy requiring therapy during the time frame of individual patient study participation.
4. Chemotherapy, radiotherapy, or immunotherapy within 4 weeks prior to Iodine (124I) Girentuximab infusion on Day 0 or continuing adverse effects (>grade 1) from such therapy.
5. Exposure to murine proteins or chimeric antibodies within the last 5 years.
6. Intercurrent medical condition that may limit patient's study participation or compliance.
7. History of autoimmune hepatitis.
8. Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study.
9. Participation in any other clinical trial involving another investigational product within 4 weeks prior to enrollment.
10. Women who are pregnant or breastfeeding.
11. Contraindication to KI intake (see package insert/Appendix VI).
12. Hyperthyroidism, or Grave's Disease.
13. Contraindication for PET/CT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of Iodine (124I) Girentuximab PET/CT scans will be compared to the threshold value of 0.70 using a two-sided exact binomial test at level 0.05. | PET/CT imaging of the kidneys will be performed 5 (±1) days (Day 4, 5, or 6) after the Iodine (124I) Girentuximab infusion.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - David Geffen School of Medicine, UCLA, Los Angeles, California
  - H. Lee Moffitt Cancer Center & Research Center, Tampa, Florida
  - Lahey Clinic, Burlington, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson, Houston, Texas